CLINICAL TRIAL: NCT00821431
Title: A Phase II Study to Compare the Effect of a Compression Device to That of a 4-layer Compression System on Subjects With Venous Leg Ulcers.
Brief Title: Compression Device Versus 4-layer Compression System
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ConvaTec Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CW-0500-05-U342
Record Dates: First submitted 2009-01-09; First posted 2009-01-13 (Estimated); Results first posted 2015-01-09 (Estimated); Last update posted 2015-01-09 (Estimated); Status verified 2015-01

CONDITIONS: Leg Ulcers
MeSH Terms: conditions — Leg Ulcer | interventions — Intermittent Pneumatic Compression Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Compression device (Experimental): The electrical compression device is operated from battery or a main adaptor. It is based upon the use of inflatable pneumatic cuffs that apply controlled compression to the foot, ankle and calf.
  Interventions: Device: Compression Device
- Profore, 4-layer bandage (Active Comparator): A high compression 4-layer bandage (Profore, Trademark of Smith and Nephew). This is a four-layer system that can be purchased either separately or as a package: a wound contact layer (Knitted viscose), a sub-compression wadding bandage, two layers of elastane bandage plus a top cohesive layer.
  Interventions: Device: Profore

INTERVENTIONS:
Device: Compression Device — Subjects randomized to the compression device regime were instructed to wear the compression device for all wakings hours for 12 weeks. The device was applied at the following pressures:
  Foot 40 mmHg, ankle 40 mmHg, mid-calf 30 mmHg, upper cuff 20 mmHg.
  Subjects were instructed to wear the Intermittent Pneumatic Compression for 2 hours per day.
  Arms: Compression device
Device: Profore — Subjects randomised to the 4-layer compression bandage regime, Profore, were to wear the bandage system for 24 hours a day and bandage applications/dressing changes were to be performed by a trained health care professional. Four different sizes of Profore were available and size selection was based on measurement of the ankle circumference of the subject on the index leg. Profore was to be used according to the instructions provided by the manufacturer described in their package insert.
  Arms: Profore, 4-layer bandage

SUMMARY:
A prospective, Phase II, stratified, randomized study to compare the safety, ulcer healing, patient compliance (concordance) and resource utilisation of a compression device with IPC mode to a Class 3(c) UK standard graduated compression regime (4- layer system) on subjects with venous leg ulcers.

ELIGIBILITY:
Inclusion Criteria:

* Subjects over 18 years, willing and able to provide written informed consent
* Subjects able to wear the compression device and the comparative regime and follow the requirements of the clinical investigation plan
* Subjects who had an ankle to brachial pressure index (ABPI) of 0.8 or greater
* Subjects who had a chronic venous leg ulcer (i.e. CEAP classification of C6 1) 2 cm2 in size or greater, who required graduated compression
* Subjects who were outpatients

Exclusion Criteria:

* Subjects with a history of skin sensitivity to any of the components of the study product, comparator product or standard dressings
* *Subjects with more than one ulcer on the test leg
* Subjects who had previously been entered into the study or a previous Amadeus study (U327, U332 or U337) or had participated in a previous clinical study within the past 3 months
* Subjects with any condition that prevented application and removal of the device without external assistance
* Subjects who had an active Deep Vein Thrombosis (DVT) or a recent DVT within the last 3 months
* Subjects who exhibited any other medical condition which, according to the Investigator, justified the subject's exclusion from the study
* Subjects who had leg sizes outside the following range:

  * Ankle - 12cm to 44cm
  * Calf - 22cm to 60cm
  * Below knee - 22cm to 68cm
* Subjects who had an index venous leg ulcer greater in size than 10cm in any one dimension
* Diabetic subjects with advanced small vessel disease
* Denotes the exclusion criterion was amended and approved by the Ethics Committees as follows:
* Amendment #1 dated 27th March 2007:

  *Diabetic subjects who, in the opinion of the investigator, were not in reasonable metabolic control or had a history of hospitalisation within the last six months for the management of blood sugar and/or diabetic subjects with advanced small vessel disease
* Amendment #2 dated 2nd August 2007:

  *Subjects who had an index venous leg ulcer greater in size than 15cm in any one dimension
* Amendment #3 dated 5th October 2007:

  * Deletion of exclusion criterion 'Subjects with more than one ulcer on the test leg' to permit inclusion of subjects with multiple ulcers on the test leg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2006-05; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathon Hopper, MD, Study Director — ConvaTec Inc.
Locations (20):
- France (2):
  - Private Practice, Neuilly-sur-Seine
  - Groupe Hospitalier Saint-Joseph, Paris
- Germany (3):
  - Hautarzt Phlebologe Allergologe, Freiburg im Breisgau
  - Private Practice, Gilching
  - Private Practice, Hamburg
- Ireland (3):
  - The Adelaide & Meath Hospital, Dublin
  - Mid-Western Regional Hospital, Limerick
  - Cork University Hospital, Wilton
- United Kingdom (12):
  - Dermatology Day Unit; Monklands Hospital, Airdrie
  - The Wilson Practice, Alton Health Centre, Alton
  - Wound Healing Research Unit; Cardiff University, Cardiff
  - Tissue Viability Consultancy, Eastbourne
  - Institute of Wound Care, The University of Hull, Hull
  - Diving Diseases Research Centre, Hyperbaric Medical Centre, Plymouth
  - University Dept of Vascular, Solihull
  - Medical Physics & Bioengineering, Southampton University Hospital, Southampton
  - Department of Vascular Surgery, Good Hope Hospital, Sutton Coldfield
  - Trowbridge Community Hospital, Trowbridge
  - Arrowe Park Hospital, Upton
  - Short Health Clinic, Willenhall

RESULTS

PARTICIPANT FLOW:
Groups:
- Compression Device: The electrical compression device is operated from battery or a main adaptor. It is based upon the use of inflatable pneumatic cuffs that apply controlled compression to the foot, ankle and calf.
  Compression Device: Subjects randomized to the compression device regime were instructed to wear the compression device for all wakings hours for 12 weeks. The device was applied at the following pressures:
  Foot 40 mmHg, ankle 40 mmHg, mid-calf 30 mmHg, upper cuff 20 mmHg.
  Subjects were instructed to wear the Intermittent Pneumatic Compression for 2 hours per day.
Period: Overall Study
Arm/Group | Compression Device | Profore, 4-layer Bandage
Started | 38 | 52
Completed | 23 | 47
Not Completed | 15 | 5
Not completed — Adverse Event | 6 | 3
Not completed — Withdrawal by Subject | 5 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 3 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Compression Device | Profore, 4-layer Bandage | Total
Number analyzed (Participants) | 38 | 52 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.9 (16.72) | 62.6 (15.41) | 61.89 (15.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 23 | 44
  Male | 17 | 29 | 46
Region of Enrollment [Number; unit: participants]
  France | 1 | 5 | 6
  Ireland | 5 | 5 | 10
  Germany | 9 | 12 | 21
  United Kingdom | 23 | 30 | 53

OUTCOME MEASURES:

1. Primary Outcome: Safety Measured by the Number of Subjects With Adverse Events (Including Any Deterioration of Ulcer)
Time Frame: 12 Weeks
Measure: Number; unit: Number of Subjects with Adverse Events
Arm/Group | Compression Device | Profore, 4-layer Bandage
Number analyzed (Participants) | 38 | 52
Number of Subjects with Adverse Events | 33 | 47

2. Secondary Outcome: Healing Measured by Number of Subjects Healed During the 12 Week Study Period
Time Frame: 12 weeks
Measure: Number; unit: Number of subjects healed
Arm/Group | Compression Device | Profore, 4-layer Bandage
Number analyzed (Participants) | 38 | 52
Number of subjects healed | 12 | 22

ADVERSE EVENTS:
Arm/Group | Compression Device | Profore, 4-layer Bandage
Serious Adverse Events (participants affected / at risk) | 0/38 | 3/52
Other Adverse Events (participants affected / at risk) | 33/38 | 47/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Compression Device (N=38) | Profore, 4-layer Bandage (N=52)
Blisters/ulcer/skin breakdown/weepy under wfr/dsg (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Prostatic Procedures (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Compression Device (N=38) | Profore, 4-layer Bandage (N=52)
Maceration (Skin and subcutaneous tissue disorders) | 18 | 13
Pain attributed to wound (Skin and subcutaneous tissue disorders) | 12 | 11
Erythema (Skin and subcutaneous tissue disorders) | 11 | 17
Eczema/worsening (Skin and subcutaneous tissue disorders) | 7 | 19
Blisters/ulcer/skin breakdown/weepy under wfr/dsg (Skin and subcutaneous tissue disorders) | 6 | 7
Oedema (Blood and lymphatic system disorders) | 6 | 3
Dry/Flaky skin under device (Skin and subcutaneous tissue disorders) | 6 | 9
Infection, Non-Study Location (Infections and infestations) | 5 | 1
Infection, Study Location (Infections and infestations) | 5 | 9
Increase in drainage/exudate (Blood and lymphatic system disorders) | 5 | 7
Pain lower leg (Vascular disorders) | 4 | 9
Wound enlarged/deteriorated (Skin and subcutaneous tissue disorders) | 3 | 7
Necrotic or sloughy wound (Skin and subcutaneous tissue disorders) | 2 | 1
Hypergranulation (Skin and subcutaneous tissue disorders) | 2 | 4
Chafing under device (Skin and subcutaneous tissue disorders) | 2 | 2
Blstrs/ulcr/skin brkdwn/weepy-diff.location (Skin and subcutaneous tissue disorders) | 2 | 0
Pain/discomf at ankle, study leg (Skin and subcutaneous tissue disorders) | 2 | 4
Pain/discomf at shin, study leg (Skin and subcutaneous tissue disorders) | 2 | 1
Pain/discomf at ankle w/irrit, study leg (Skin and subcutaneous tissue disorders) | 2 | 0
Headache (General disorders) | 2 | 0
Cellulitis (Infections and infestations) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No